

### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

Phase I/II Trial of Encorafenib, Cetuximab, and Nivolumab in Microsatellite Stable BRAFV600E Metastatic Colorectal Cancer (BMS-MDACC CA209-8P6/ARRAY IST-818-101X) 2018-0993

| Subtitle: BMS-MDACC CA209-8P6/ARRAY IST-818-101X | | |
|---|---|---|
| Study Chair: | Van K. Mor | ris |
| Participant's Name | | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

### STUDY SUMMARY

The goal of this clinical research study is to learn if the combination of encorafenib, cetuximab, and nivolumab can help to control colorectal cancer that is metastatic (has spread). The safety of this drug combination will also be studied.

This is an investigational study. Cetuximab is FDA approved and commercially available for the treatment of colorectal cancer. Encorafenib and nivolumab are FDA approved for the treatment of other types of cancer, but not this type of colorectal cancer. The use of all 3 study drugs in combination is investigational. The study doctor can explain how the study drugs are designed to work.

Taking the study drug may help to control the disease. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side

effects, potential expenses, and time commitment. If you take part in this study, you may experience side effects (including rash, fatigue, abdominal pain, nausea and/or vomiting, and changes in body salts), costs due to travel to and from MD Anderson, and/or hospitalization if the side effects become severe or unsafe. You should also be aware that this is the first study using this drug combination in humans.

Currently, the standard-of-care for patients with this type of colorectal cancer here would be chemotherapy in combination with a drug like cetuximab that has been shown to prolong survival in other research studies. By receiving the treatment on this research study, you are passing on the opportunity to receive standard therapies. However, these therapies (chemotherapy) may be available for you, based on the opinion and recommendation of your doctor, to receive should the treatment on the clinical trial not work.

You can read a list of potential side effects below in the Possible Risks section of this consent.

You may continue receiving the study drugs for as long as the doctor thinks it is in your best interest. Sometimes with a drug like nivolumab, tumors may get slightly larger before they start to get smaller. In this event, at the opinion of your doctor, you may be allowed to continue on treatment as part of this research study until tumors increase further in size at a later point in time.

Nivolumab and encorafenib will be provided at no cost to you while you are on study. You and/or your insurance provider will be responsible for the costs of cetuximab.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive other investigational therapy, if available. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

### 1. STUDY DETAILS

### Screening Tests

Signing this informed consent form does not mean that you will be able to take part in this study. Within 28 days before your first dose of study drug you will have screening tests to help the doctor decide if you are eligible:

- You will have a physical exam. This will include a skin exam by the study doctor.
- Blood (about 3 teaspoons) will be drawn for routine tests. If you can become pregnant, this blood or a urine sample will also be used for a pregnancy test. To take part in this study, you must not be pregnant.
- You will have 3 EKGs in a row (triplicate EKGs) to check your heart function.
- You will have an eye exam performed by an eye doctor.
- You will have a CT scan or MRI to check the status of the disease.
- If it is available, leftover tumor tissue from a previous procedure will be collected for biomarker testing.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other options will be discussed with you.

Up to 48 participants will be enrolled in this study. All will take part at MD Anderson.

### Study Drug Administration

If you are found to be eligible to take part in this study, you will receive the study drugs in 28-day cycles:

- You will take encorafenib by mouth at about the same time every day with about a cup (8 ounces) of water. You can take it with or without food.
- You will receive cetuximab by vein over about 1 hour on Days 1 and 15 of each cycle (every 2 weeks).
- You will receive nivolumab by vein over about 30 minutes on Day 1 of each cycle (every 4 weeks).

On days that you receive drugs by vein, you must take your dose of encorafenib at least 1 hour before you receive any other drugs.

If you vomit at any time after taking encorafenib, you should not take another dose.

You will receive a diary to record when you take encorafenib each time. You will also write the dose taken and if any doses were missed and the reason for the missed dose. You will be instructed to return unused encorafenib and the patient diary to the site at the end of each cycle.

You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your active participation in this study will be over after the follow-up visit.

### Study Visits

You will have study visits on Days 1 and 15 of every cycle. At each study visit:

- You will have a physical exam. Every 2 months, this will include a skin exam.
- Blood (about 2-4 teaspoons) will be drawn for routine tests. At some of these visits, this will also include biomarker testing.

Additionally, some tests and procedures will only be performed at certain visits:

- On Day 1 of each cycle, if you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.
- On Day 15 of Cycle 1, and then on Day 1 of every odd-numbered cycle (3, 5, and so on), you will have an EKG.
- On Day 1 of every even-numbered cycle (2, 4, and so on), you will have an eye exam.
- On Day 1 of every odd-numbered cycle, you will have a CT scan or MRI to check the status of the disease.

At any time during the study, you may have some of the above tests repeated if the doctor thinks they are needed for your safety. The study doctor will tell you if you need to have any of these tests repeated.

# **End-of-Dosing Visit**

As soon as possible after your last dose of study drugs:

- You will have a physical exam, including a skin exam.
- Blood (about 2 teaspoons) will be drawn for routine tests.
- You will have an eye exam.
- If the disease appears to have gotten worse, blood (about 2 teaspoons) will be drawn for biomarker testing.

### Follow-Up

About 30 and 100 days after the end-of-dosing visit:

- You will have a physical exam, including a skin exam.
- Blood (about 2 teaspoons) will be drawn for routine tests.
- If you had a side effect related to your eye at the end-of-dosing visit, you will have an eye exam at the 30-day follow-up visit.
- If you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

If you stopped receiving the study drugs for reasons other than the disease getting worse, you will have CT scans or MRIs every 8 weeks for up to 2 years after your last dose.

About 3 months after your end-of-dosing visit and then every 3 months until the study is over, you will be called by the study staff and asked how you are doing and if you have taken any other anticancer treatments. Each call should last about 10-15 minutes.

### Other Information

- During the study, you will not be allowed to receive other treatments for cancer including chemotherapy, immunotherapy, hormonal therapy, radiation therapy, and/or biologic therapy.
- You should tell the study staff about any over-the-counter drugs, herbal supplements, vitamins, and prescription drugs you may be taking while you are on study.
- You should not have any vaccinations while you are taking the study drug-
- You must avoid eating grapefruit, pomegranates, star fruits, Seville oranges, or products containing the juice of each during the entire study. You should not eat or drink these starting at least 7 days before your first dose. Regular orange juice is allowed.

### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drug/procedures.

Nivolumab, cetuximab, and encorafenib may each cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become lifethreatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

### Nivolumab Side Effects

# Common (occurring in more than 20% of patients)

- fatigue/lack of energy
- headache
- fever
- skin rash
- itching
- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)
- high blood levels of fat (possible heart disease and/or stroke)

- high blood sugar (possible diabetes)
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- abdominal pain
- diarrhea
- loss of appetite
- nausea
- constipation
- abnormal digestive blood test (possible inflammation of the pancreas)

- low blood cell counts (red, white, platelets)
- abnormal liver test (possible liver damage and/or yellowing of the skin and/or eyes)
- pain
- abnormal kidney test (possible kidney damage)
- weakness
- difficulty breathing
- cough
- infection

# Occasional (occurring in 3-20% of patients)

- swelling (arm/leg)
- dizziness
- skin redness
- patches of skin color loss
- overactive thyroid gland (possible weight loss, heart rate changes, and/or sweating)
- inflammation of the thyroid gland (possible tenderness in the neck)
- vomiting
- inflammation of the intestines
- hole in the intestines (possibly leaking contents into the abdomen)

- mouth blisters/sores (possibly difficulty swallowing)
- abnormal blood test (possible pancreas damage)
- nerve damage (possible numbness, pain, and/or loss of motor/sensory function)
- inflammation of nerves (possible pain and/or loss of motor or sensory function)
- peripheral nerve palsy (weakness, numbness, tingling)
- muscle damage causing weakness

- joint disease
- build-up of fluid around the lungs
- lung inflammation (possible difficulty breathing)
- stuffy nose
- immune reaction (possible organ damage)
- immune system disease (possible dry mouth/eyes, fatigue, joint pain, and/or organ failure)
- infusion reaction (possible chills and/or hives)

If you have a stem cell transplant from a donor before or after you receive nivolumab, you may have an increased risk of complications, such as severe graft-versus-host disease (when transplanted donor tissue attacks the recipient's organs such as skin, liver, and/or intestines) and/or clotting of blood within the liver. Deaths have been reported in patients who received stem cell transplant from a donor before or after nivolumab therapy. If you decide to receive a stem cell transplant from a donor, please tell your transplant doctor that you received nivolumab in the past.

# Rare but serious (occurring in fewer than 3% of patients)

- blood vessel inflammation (possible bleeding and/or bruising)
- heart inflammation
- brain inflammation (possible paralysis and/or coma)
- damage to the nervous system (causing numbness and/or paralysis)
- paralysis of the nerves controlling the head and neck
- skin blisters

- hormonal deficiency that affects the body's ability to control blood pressure and react to stress
- inflammation of the pancreas (possible abdominal pain)
- liver damage (possibly due to blood clots)
- paralysis (face)
- uncontrolled movements

- blockage in the lung (possible pain and/or shortness of breath)
- multi-organ disease causing lesions, most often in the lungs (sarcoidosis)
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)
- Vogt Koyanagi Harada syndrome -pigmented tissue

| <ul> <li>diabetes</li> <li>kidney failure</li> <li>breakdown of muscle</li> <li>tissue (possibly kidney</li> </ul> |
|---|
|---|

### Frequency unknown

| <ul> <li>migraine</li> <li>very severe blistering skin<br/>disease (loss of large<br/>portion of skin and/or<br/>ulcers of the skin and<br/>digestive tract)</li> </ul> | <ul> <li>hand-foot syndrome<br/>(palms of hands/soles<br/>of feet having pain,<br/>swelling, and<br/>blistering)</li> </ul> | weight loss |
|---|---|---|
|---|---|---|

You may need to take drugs to reduce inflammation while taking nivolumab. Long-term use of these drugs may increase your risk of infection. These infections may occur anywhere and may be fatal. Treatment with antibiotic or antifungal drugs may be required to treat these infections.

The study drug works by boosting the immune system. This may cause unknown side effects resulting from your immune system attacking your organs. This may cause inflammation and inflammation-related side effects in any organ or tissue.

Nivolumab may cause serious side effects that affect your immune system. Some of these side effects start as inflammation in different areas of the body like the skin, hormone glands, pancreas, or appendix. Tell the study staff right away if you have diarrhea, nausea, vomiting, blurred vision, dizziness, fainting, or you are feeling cold all the time.

If you had an organ transplant, nivolumab may increase your risk for the transplant to be rejected by your body.

# Cetuximab Side Effects

# Common (occurring in more than 20% of patients)

| • fever | diarrhea | Pain |
|---|---|---|
| difficulty sleeping | <ul> <li>constipation</li> </ul> | • pain |
| headache | <ul> <li>abdominal pain</li> </ul> | <ul><li>weakness</li></ul> |
| <ul> <li>fatigue/lack of energy</li> </ul> | <ul> <li>dehydration</li> </ul> | (possible liver damage) |
| heart attack | <ul><li>weight loss</li></ul> | <ul> <li>abnormal liver tests</li> </ul> |

- skin rash (possibly acnelike), peeling, and/or itching
- dry skin
- nail changes
- low blood levels of magnesium (possible weakness and/or seizures)
- mouth blisters/sores (possible difficulty swallowing)
- vomiting
- nausea
- loss of appetite
- low white blood cell count
- nerve damage (loss of sensory function)
- difficulty breathing
- cough
- sore throat
- infection
- severe rash at the site of previous radiation
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)

# Occasional (occurring in 3-20% of patients)

- confusion
- depression
- anxiety
- chills/shivering
- skin sores
- hair loss (partial or total)
- hand-foot syndrome (palms of hands/soles of feet having pain, swelling, and blistering)
- low blood levels of calcium and/or potassium (possible weakness and/or cramping)
- dry mouth
- abnormal taste
- upset stomach

- painful red eyes
- immune reaction
- infusion reaction (possible chills and/or hives)
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)

# Frequency unknown but occurring in 1-10% of patients

hair growth

# Rare but serious (occurring in fewer than 3% of patients)

- heart attack
- stoppage of heart and lung function
- decreased blood supply to the heart
- low blood pressure (possible dizziness/fainting)
- irregular heartbeat
- inflammation of the membranes around the

- shock
- loss of consciousness
- large skin blisters
- very severe blistering skin disease (with ulcers of the skin and digestive tract)
- very severe blistering skin disease (loss of large portion of skin)

- eye ulcer
- kidney failure
- lung inflammation (possible difficulty breathing)
- difficulty breathing due to narrowing of the airways
- blockage in the lung (possible pain, shortness of breath,

| spinal cord and brain<br>(possible headache<br>and/or coma) | <ul> <li>changes in body salts<br/>such as sodium<br/>and/or potassium<br/>(possible fatigue<br/>and/or weakness)</li> </ul> | and/or failure to<br>breathe) |
|---|---|---|
|---|---|---|

### **Encorafenib Side Effects**

# Common (occurring in more than 20% of patients)

- headache
- fatigue
- thickening of external part of the skin
- hand-foot syndrome (palms of hands/soles of feet having pain, swelling, and blistering)
- dry itching skin
- skin rash (including an acne-like rash)
- loss of hair (partial or total)
- high blood sugar (possible diabetes)
- nausea/vomiting
- abdominal pain
- constipation
- abnormal liver tests (possible liver damage)
- low red blood cell count
- abnormal kidney tests (possible kidney damage)
- pain

# Occasional (occurring in 3-20% of patients)

- fever
- dizziness
- abnormal taste
- difficulty sleeping
- skin redness
- pre-cancerous skin lesion
- inflammation of the fatty layer under the skin
- skin tags
- new moles or changes in existing moles
- low blood levels of sodium (possible headache, confusion, seizures, and/or coma)

- high blood levels of magnesium (possible abnormal muscle function and/or blood pressure)
- indigestion
- loss of appetite
- bleeding or blood/bright red blood in the stool
- inflammation of the pancreas (possible abdominal pain)

- low white blood cells
- bleeding
- muscle spasm
- weakness (facial muscles)
- nerve damage (possible numbness, pain, and/or loss of motor function)
- inflammation inside the eye (possible vision problems)
- allergic reaction

# Rare but serious (occurring in fewer than 3% of patients)

abnormal EKG

Encorafenib may cause you to develop a new type of melanoma, basal cell carcinoma, and squamous cell carcinoma (a type of skin cancer).

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

### Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

During the **eye exam**, your pupils will be dilated with eye drops to allow a good view of the back of the eye. This will result in some blurred vision lasting for a few hours. You will not be able to drive during this time.

**EKGs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

During the **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.

CT scans send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study. Only the study staff will have access to study data.

This study may involve unpredictable risks to the participants.

### **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. If you are sexually active, you must use birth control while on study and for 100 days after your last dose of study drug.

Birth Control Specifications: If you can become pregnant or father a child, you must use 2 forms of acceptable highly effective birth control, one of which must be a barrier method (condom, diaphragm, or cervical/vault cap). Hormonal methods (like birth control pills) can only be used in combination with another highly effective form of birth control.

Highly effective forms of birth control include:

- Birth control pills, patch, injections, or implants
- Intrauterine device or system (IUD or IUS)
- Barrier methods with spermicide
- Surgical sterilization (bilateral oopherectomy with or without hysterectomy, tubal ligation, or vasectomy) of you or your partner at least 6 weeks before taking the study drugs.

Males: Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away.

Getting pregnant will result in your removal from this study.

#### OPTIONAL PROCEDURES FOR THE STUDY

**Optional Procedure #1:** If you agree, you will have a core needle biopsy before you start study treatment, before day 1 of cycle 2 of treatment, and/or if at any point the disease gets worse. This will be done to help researchers understand why the study drugs may not have worked or stopped working.

There are no benefits to you for taking part in the optional procedure. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedure.

### **Optional Procedure Risks:**

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

### CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1**: Do you agree to have tumor biopsies?

YES NO

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson, Bristol-Myers Squibb, or Pfizer for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

### **Additional Information**

- 4. You may ask the study chair (Dr. Van K. Morris, at 713-792-2828) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. It may be harmful to suddenly stop receiving the study drugs. If you withdraw from this study, you can still choose to be treated at MD Anderson. You may be asked to continue to allow the study staff to collect information from your medical record about your routine care.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Bristol-Myers Squibb, Pfizer, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, including the results of all of your standard tests performed as part of this research, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: Bristol-Myers Squibb and Pfizer.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

#### **Future Research**

Your personal information and/or samples are being collected as part of this study. These data and/or samples may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

Before being shared for future research, every effort will be made to remove your identifying information from any data and/or samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or samples are used for future research. If this research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

### **Genetic Research**

Samples collected from you as part of this study will be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment.

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

### Conflict of Interest

Outside relationships are disclosed to and approved by the Conflict of Interest Committee, which reviews these relationships for compliance with institutional policy. This review helps the IRB to assure that financial relationships do not have an impact on the conduct of this study. The following members of the study staff have

disclosed compensation from the funding source(s) of this study:

- Van Morris (Principal Investigator)
- Scott Kopetz, Michael Overman, and Kanwal Raghav (Co- Investigators)

## Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Bristol-Myers Squibb and Pfizer, who are sponsors or supporters of this study, and/or any future sponsors/supporters of the study
  - Any future sponsors and/or licensees of the study technology
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

Informed consent documents will remain in the electronic medical record indefinitely (without a set end date) as part of each participant's medical record. De-identified data as part of the study database is password protected and locked at the time that the study ends, and will be accessible only to the study doctor.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.

Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.

- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the

| consent form for this study, or have had it read to me. I have had a c about it, ask questions, and talk about it with others as needed. I give permission to enroll me on this study. By signing this consent form, I any of my legal rights. I will be given a signed copy of this consent d | e the study chair<br>I am not giving up |
|---|---|
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be performed | under this protocol. |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | DATE |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his o representative, using language that is understandable and appropria have fully informed this participant of the nature of this study and its pand risks and that the participant understood this explanation. | te. I believe that I |
| PERSON OBTAINING CONSENT | DATE |

PRINTED NAME OF PERSON OBTAINING CONSENT

| <u>TRANSLATOR</u> | | |
|---|---|---|
| I have translated the above in subtractions) into | nformed consent as written (without addition<br>and assisted the | |
| , (N | lame of Language) | |
| obtaining and providing cons<br>consent process for this parti | ent by translating all questions and respons<br>cipant. | es during the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| | ranslator was a member of the research tea<br>Islator, must sign the witness line.) | ım. (If checked |